CLINICAL TRIAL: NCT05652478
Title: A Phase 2 Randomized Cross-Over Design Study of the Early Metabolic Effects of Dolutegravir or Tenofovir Alafenamide in Healthy Volunteers
Brief Title: Early Metabolic Effects of Dolutegravir or Tenofovir Alefenamide in Healthy Volunteers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 10000906; 000906-I
Record Dates: First submitted 2022-12-10; First posted 2022-12-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-13

CONDITIONS: Healthy Volunteer; Weight Gain; Metabolic Effects; Integrase Strand Transfer Inhibitors
Keywords: Metabolism; HIV; Integrase Strand Transfer Inhibitors
MeSH Terms: conditions — Weight Gain | interventions — tenofovir alafenamide; dolutegravir

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolutegravir (Active Comparator): 50mg one tablet orally once daily for 8 days.
  Interventions: Drug: Dolutegravir
- Tenofovir alafenamide (Active Comparator): 25mg one tablet orally once a day for 8 days.
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Tenofovir alafenamide — 25mg tenofovir alafenamide (TAF) one tablet orally once a day for 8 days.
  Arms: Tenofovir alafenamide
Drug: Dolutegravir — 50mg dolutegravir (DTG) one tablet orally once daily for 8 days.
  Arms: Dolutegravir

SUMMARY:
Background:

People with HIV take drugs to keep the amount of virus in their body low. One type of these drugs, called integrase strand transfer inhibitors (INSTIs), can cause weight gain over time. Weight gain can cause diabetes, heart disease, and other serious issues. Researchers want to understand how INSTIs cause weight changes.

Objective:

To see how a common INSTI, dolutegravir (DTG), affects how the body uses energy. DTG will be compared with a non-INSTI drug, tenofovir alafenamide (TAF).

Eligibility:

Healthy people aged 18 to 55.

Design:

Participants will be screened. They will have a physical exam and blood tests. They will have a nutritional assessment and tests of their heart function.

Participants will have 2 inpatient stays at the clinic. Each stay will be for 11 nights, with a 3-week break between.

Both DTG and TAF are gel caps swallowed once per day by mouth. Participants will take 1 drug for 8 days during each stay.

Participants will have tests to see how their body uses energy:

They will spend 23 continuous hours in a special room that measures how much oxygen they breathe in and how much carbon dioxide they breathe out. They will do this a total of 6 times.

They will have a DEXA (dual-energy X-ray absorptiometry). DEXA is a kind of X-ray that measures body fat and bone density.

They will lie on a table. Electrodes will be placed on their hands and feet to measure body fat and lean body mass.

They will stand still on a platform for about 30 seconds. High-resolution laser cameras will scan their bodies.

DETAILED DESCRIPTION:
Study Description:

Integrase strand transfer inhibitors (INSTIs) are a class of antiretroviral (ARV) drugs currently included in first-line therapy to treat HIV infection. Several observational trials have shown that one side effect of this class of ARVs is involuntary weight gain. How these drugs cause weight gain is unknown. In addition, these marketed drugs are formulated in combination with the nucleotide reverse transcriptase inhibitor (NRTI) tenofovir alafenamide (TAF), which may also independently contribute to weight gain, as compared to the older formulation of tenofovir disoproxil fumarate (TDF). To better understand the effects of INSTIs and TAF on metabolism, participants will be randomized 1:1 to either the INSTI dolutegravir (DTG) or TAF. Participants will be admitted to the Metabolic Unit of the NIH CC, undergo an initial baseline evaluation over 3 days, followed by an 8-day period during which they will take either drug (TAF or DTG) once daily. Following an 18-day washout period at home, participants will then be readmitted to the Metabolic Unit and assigned to the other drug, which they will follow for another 8 days. Throughout the study, participants will be assessed for metabolic processes, including 24-hour energy expenditure via metabolic chamber.

Primary Objective:

To determine if TAF or DTG induce changes in 24-hour energy expenditure and 24-hour respiratory quotient (RQ).

Secondary Objectives:

1. To determine if baseline demographic (eg, age, sex, or weight) or laboratory characteristics (eg, free thyroxine [T4], thyroid-stimulating hormone [TSH], cortisol, or other hormones) are associated with changes in 24-hour energy expenditure.
2. To determine if there is a correlation between steady-state pharmacokinetics of TAF or DTG and changes in 24-hour energy expenditure or caloric intake.

Exploratory Objective:

Evaluation of microbiota in vaginal, oral, and rectal mucosa, including potential reactivation of human endogenous retroviruses (HERVs) at start and the end of each treatment period (TAF and DTG).

Primary Endpoint:

Change in 24-hour energy expenditure and 24-hour RQ from baseline to day 1 and day 8 of ARV therapy with each drug.

Secondary Endpoints:

1. Relationship between demographic data or baseline laboratory values and changes in energy expenditure or caloric intake.
2. Relationship between pharmacokinetic parameters for TAF and DTG and changes in energy expenditure or caloric intake.

Exploratory Endpoint:

Potential changes in microbiome composition and HERVs reactivation after treatment periods with TAF or DTG.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged 18 to 55 years.
* Able to provide informed consent.
* Willing and able to stay in the whole-room indirect calorimetry suite on 6 occasions.
* Willing to reside on the metabolic unit in the Clinical Center for 2 stays of 11 consecutive days over the course of 5 weeks.
* Willing to allow samples and data to be stored and shared for future research.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Current infection with HIV or hepatitis A, B, or C.
* Body mass index (BMI) <18.5 kg/m^2 or >30.0 kg/m^2.
* Weight change >5% in the past 6 months or a trained athlete.
* History of or current cardiovascular disease such as congestive heart failure, heart block, or clinically relevant abnormal ECG as determined by investigators.
* History of or current liver disease or alanine transaminase serum level >2x upper limit of normal.
* History of or current kidney disease or renal insufficiency, or estimated creatinine clearance <=50 mL/min (Modification of Diet in Renal Disease equation).
* Current cancer or history of cancer within 5 years of screening, with the exception of squamous cell carcinoma or basal cell carcinoma that is localized and does not require systemic therapy.
* History of bariatric surgery.
* Diabetes mellitus.
* Fasting serum glucose >126 mg/dL.
* History of or current hypo- or hyper-thyroid or abnormal TSH, except minor deviations deemed to be of no clinical significance by the investigator.
* History of or current asthma or chronic obstructive pulmonary disease.
* History of or current glaucoma.
* Psychological conditions by self-report, such as (but not limited to) claustrophobia, clinical depression, bipolar disorders, that would be incompatible with safe and successful participation in this study.
* Pregnancy or within 1 year post-partum.
* Experiences irregular menstrual cycles.
* Breastfeeding.
* Blood pressure >140/90 mm Hg or current antihypertensive therapy.
* Anemia, defined as hemoglobin <13 g/dL (males) or <12 g/dL (females).
* History of illicit drug, opioid, or alcohol abuse within the last 5 years; current use of illicit drugs or opioids (by history) or excessive alcohol (CAGE assessment score >=2).
* Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism.
* Current use of the following prescription or over-the-counter medications and supplements:

  * Carbamazepine
  * Oxcarbazepine
  * Phenobarbital
  * Phenytoin
  * Primidone
  * Rifabutin
  * Rifampin
  * Rifapentine
  * St. John's wort (Hypericum perforatum)
  * Cation-containing antacids or laxatives
  * Sucralfate
  * Buffered medications
  * Oral calcium, iron, magnesium, or zinc supplements, including multivitamins containing these polyvalent cations
  * Dalfampridine
  * Metformin
  * Dofetilide
  * Thyroid medications
  * Corticosteroids
  * Weight loss medications, including prescription drugs (eg, semaglutide and tirzepatide) and over-the-counter diet pills
  * Hormone medications for any indication
* Use of tenofovir alafenamide (Descovy) or tenofovir disoproxil fumerate (Truvada) for the purpose of HIV PrEP within the past 6 months.
* Any history of exposure to cabotegravir (eg, as HIV PrEP or as a participant in research study for this drug).
* Current use of nonprescriptive medications that may have interactions with study drugs as determined by the investigators.
* History of adverse or allergic reactions to the study drugs.
* Daily caffeine intake >500 mg (about 4 cups of coffee)
* Current smoker or user of tobacco products.
* Participants with dietary allergies, intolerances, or eating patterns that would preclude them from consuming controlled metabolic meals.
* Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour energy expenditure and 24-hour RQ from baseline to day 1 and day 8 of ARV therapy with each drug | Baseline to day 1 and Day 8 of ARV therapy for drug regimen.
  To determine if TAF or DTG induce changes in 24-hour energy expenditure and 24-hour respiratory quotient (RQ)

SECONDARY OUTCOMES:
Relationship between demographic data or baseline laboratory values and changes in energy expenditure or caloric intake | Throughout study
  To determine if baseline demographic or laboratory characteristics are associated with changes in 24-hour energy expenditure.
Relationship between pharmacokinetic parameters for TAF and DTG and changes in energy expenditure or caloric intake. | Days 10 and 38
  To determine if there is a correlation between steady-state pharmacokinetics of TAF, or DTG and changes in 24-hour energy expenditure or caloric intake.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Epling, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We have no plans to share data with anyone outside of the study team for this pilot study.

REFERENCES:
- [Background] Squires K, Kityo C, Hodder S, Johnson M, Voronin E, Hagins D, Avihingsanon A, Koenig E, Jiang S, White K, Cheng A, Szwarcberg J, Cao H. Integrase inhibitor versus protease inhibitor based regimen for HIV-1 infected women (WAVES): a randomised, controlled, double-blind, phase 3 study. Lancet HIV. 2016 Sep;3(9):e410-e420. doi: 10.1016/S2352-3018(16)30016-9. Epub 2016 May 27. PMID 27562742
- [Background] Molina JM, Clotet B, van Lunzen J, Lazzarin A, Cavassini M, Henry K, Kulagin V, Givens N, de Oliveira CF, Brennan C; FLAMINGO study team. Once-daily dolutegravir versus darunavir plus ritonavir for treatment-naive adults with HIV-1 infection (FLAMINGO): 96 week results from a randomised, open-label, phase 3b study. Lancet HIV. 2015 Apr;2(4):e127-36. doi: 10.1016/S2352-3018(15)00027-2. Epub 2015 Mar 10. PMID 26424673
- [Background] Lennox JL, Landovitz RJ, Ribaudo HJ, Ofotokun I, Na LH, Godfrey C, Kuritzkes DR, Sagar M, Brown TT, Cohn SE, McComsey GA, Aweeka F, Fichtenbaum CJ, Presti RM, Koletar SL, Haas DW, Patterson KB, Benson CA, Baugh BP, Leavitt RY, Rooney JF, Seekins D, Currier JS; ACTG A5257 Team. Efficacy and tolerability of 3 nonnucleoside reverse transcriptase inhibitor-sparing antiretroviral regimens for treatment-naive volunteers infected with HIV-1: a randomized, controlled equivalence trial. Ann Intern Med. 2014 Oct 7;161(7):461-71. doi: 10.7326/M14-1084. PMID 25285539
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000906-I.html